CLINICAL TRIAL: NCT05341024
Title: Effect of Pelvic Floor Muscles Training on Symptoms, Bother and Amount of Stress Urinary Incontinence in Female CrossFit and Functional Fitness Exercisers. An Assessor Blinded Randomized Controlled Trial
Brief Title: Pelvic Floor Muscle Training in Female CrossFit and Functional Fitness Exercisers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Kari Bø, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLS2022
Record Dates: First submitted 2022-04-04; First posted 2022-04-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor Disorders; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 16 weeks home-based PFM training program with weekly follow-up by a physiotherapist
  Interventions: Other: Pelvic Floor Muscle Training in female CrossFit and functional fitness exercisers
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Pelvic Floor Muscle Training in female CrossFit and functional fitness exercisers — The intervention will consist of a home-based PFM training program with weekly follow-up by phone by a physiotherapist. Before commencing PFM training, the participants in the intervention group will have an individual session with a physiotherapist including thorough teaching on how to perform a correct PFM contraction (clinical exams of pelvic floor muscle function by observation and vaginal digital palpation) and instructions on how to perform the training program. The program consists of 3 sets of 8-12 maximum contractions per day. An electronic app (Athlete monitoring) will be used to assess adherence to the program. The participants will be asked to register their training sessions in a personal account. A reminder to adhere to the program will be sent by phone. The training period will be 16 weeks and the exercises will take approximately 10 minutes per day to perform.
  Arms: Intervention Group

SUMMARY:
There is a high prevalence of urinary incontinence (UI) among female athletes and exercisers, especially in sports including high impact activities and heavy weightlifting. CrossFit and functional fitness is a popular exercise form, including a combination of heavy lifting and high impact activities at high intensities. In several recent studies, high prevalence rates of UI have been reported among female CrossFit/functional fitness exercisers. UI is defined as "the complaint of involuntary loss of urine". Stress urinary incontinence (SUI) is the most common type of UI and is defined as "the complaint of involuntary loss of urine on effort or physical exertion (e.g. sporting activities), or or sneezing or coughing". Urinary leakage during sport activities may affect athletes' and exercisers' performance, cause bother, frustration and embarrassment and furthermore lead to avoidance and cessation of sport activities. Pelvic floor muscle (PFM) training is highly effective in treating SUI in the general female population. However, evidence of the effect of PFM training in exercisers participating in high impact and heavy weightlifting activities is sparse.

The purpose of this assessor-blinded randomized controlled trial (RCT) is to assess the effect of PFM training on symptoms, bother and amount of SUI in female CrossFit/functional fitness exercisers.

DETAILED DESCRIPTION:
BACKGROUND:

Physical activity and exercise have well-known beneficial effects on several physical and psychological health outcomes. However, it has been proposed that regular participation in physical activity and exercise may lead to greater risk of developing pelvic floor dysfunctions (PFD) in women. The pelvic floor consists of muscles, fascia and ligaments and forms a hammock-like support at the base of the abdomino-pelvic cavity. The function of the pelvic floor is to provide support to the pelvic organs (the bladder, urethra, vagina, uterus and rectum) and to counteract all increases in intra-abdominal pressure and ground reactions forces during daily activities. Additionally, the pelvic floor facilitates intercourse, vaginal birth, storage of stool and urine and voluntary defecation and urination. A dysfunctional pelvic floor can lead to urinary and anal incontinence, pelvic organ prolapse, sexual problems and chronic pain syndromes. UI is the most common PFD, defined as "the complaint of involuntary loss of urine". SUI, urgency urinary incontinence (UUI) and mixed urinary incontinence (MUI) are common subtypes of UI. In women, SUI accounts for approximately half of all incontinence types and is defined as "the complaint of involuntary loss of urine on effort or physical exertion (e.g. sporting activities), or on sneezing or coughing". UUI is defined as the "complaint of involuntary loss of urine associated with urgency" and MUI as "complaints of both stress and urgency urinary incontinence".

High prevalence rates of UI among both parous and nulliparous female athletes and exercisers have been reported in several cross-sectional studies. The prevalence rates varies between 0-80% with the highest prevalence found in high impact sports such as trampoline jumping, gymnastics and strengths sports with high increases in intraabdominal pressure (e.g. powerlifting). CrossFit and functional fitness, which are trending exercise forms, includes a combination of heavy lifting and high impact activities at high intensities. High prevalence of UI among CrossFit/functional fitness exercisers has been reported in several recent cross-sectional studies, ranging from 41-84%. Leakage during sport and exercise may affect performance and cause bother, frustration and embarrassment, and may further lead to avoidance or cessation of sport and exercise.

To date, there is level 1 evidence and grade A recommendation for PFM training alone to be first line treatment for SUI, MUI and pelvic organ prolapse in the general female population. In addition, PFM training is highly effective as primary prevention; pregnant continent women who exercise the PFM are at 62% less risk of UI in late pregnancy and 29% less risk of UI 3-6 months postpartum. Evidence of the effect of PFM training in athletes or strenuous exercisers is sparse.

In one study on female soldiers and two small case series in female athletes and exercisers, PFM training led to reduced symptoms of UI. However, none of these studies included a non-treated control group and the internal validity is therefore low. To our knowledge, only one RCT has assessed effects of PFM training on SUI in athletes. Female volleyball players (n=16) who followed a PFM training program had significant improvements of SUI compared to a control group (n=16).

Based on today's knowledge we do not know whether PFM training is effective in strenuous exposed to excessive impact and increases in intraabdominal pressure during CrossFit- and functional fitness activities. Given the high impact on the pelvic floor in these exercisers, it is presumed that they need much better pelvic floor muscle function than non-exercisers. On the other hand, these exercisers may be motivated for regular training. Strength training of the PFM, if proven effective, may be easily incorporated in their basic training regimens both as prevention and treatment strategies of SUI.

AIMS:

The aim of this RCT is to assess the effect of PFM training on symptoms, bother and amount of SUI among female CrossFit and functional fitness exercisers.

STUDY DESIGN AND METHODS:

To recruit participants, we will contact CrossFit boxes and functional fitness clubs in or near Oslo. Social media platforms (such as Facebook, Instagram) will also be used. The study is an assessor-blinded RCT evaluating the effect of PFM training on SUI in CrossFit and functional fitness exercisers. At baseline, a pelvic floor muscle assessment (resting pressure, strength and endurance) will be performed of all participants. In addition, the participants will respond to an electronic questionnaire, measuring self-reported symptoms of UI and bother. The participants will be randomly assigned to either a PFM training group (EG) or a control group (CG) with no intervention. The intervention consists of a daily home-based PFM training program with weekly follow-up by a physiotherapist. After a 16-week intervention period, all participants will perform a post-test including the same previous mentioned outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* ≥ 6 months of consistent participation in CrossFit or functional fitness training
* Participating in ≥ 3 sessions of cross-fit training per week
* Self-reported SUI and a total score on ICIQ-UI-SF of ≥ 3. A change of the ICIQ-UI-SF score of 2.5 has been identified to be the minimal important difference (MID) and 1.58 as between-treatment MID (Nystrom et al., 2015).
* No musculoskeletal injuries for the past 6 months with negative effect on training participation

Exclusion Criteria:

* Ongoing pregnancy, or planning to get pregnant during the intervention period
* History of hysterectomy or pelvic surgery to correct UI or POP
* History of musculoskeletal injuries for the past 6 months with negative effect on training participation
* Parous women who are ≤12 months post-partum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF) | Change in total score from baseline at four months
  A reliable and valid questionnaire assessing self-reported prevalence, amount of leakage, bother and type of UI. A change in ICIQ-UI-SF score of 1.58 points will be considered as between-treatment minimum important difference.

SECONDARY OUTCOMES:
Pelvic Floor Muscle Resting Pressure | Change in pressure value from baseline at four months
  Measurement of vaginal resting pressure will be measured with manometry. A high precision pressure transducer connected to a vaginal balloon catheter (Camtech AS, Sandvika Norway) will be used. The method has demonstrated good intra-observer reliability (intraclass correlation coefficient: >90). Vaginal resting pressure will be recorded in cmH2O.
Pelvic Floor Muscle Strength | Change in pressure value from baseline at four months
  We will use manometry to assess pressure rise generated during a maximum voluntary contraction of the PFM (PFM strength). A high precision pressure transducer connected to a vaginal balloon catheter (Camtech AS, Sandvika Norway) will be used. The method has demonstrated good intra-observer reliability (intraclass correlation coefficient: >90). Average peak pressure from 3 different PFM maximum voluntary contraction will be used to report PFM strength, recorded in cmH2O.
Pelvic Floor Muscle Endurance | Change in pressure value from baseline at four months
  We will use manometry to assess the participants ability to perform a 10 seconds sustained PFM contraction (PFM endurance). A high precision pressure transducer connected to a vaginal balloon catheter (Camtech AS, Sandvika Norway) will be used. The method has demonstrated good intra-observer reliability (intraclass correlation coefficient: >90). PFM endurance will be reported as the area under the pressure curve in cmH2O multiplied by the duration of the contraction (10 s).
Self-Efficacy Scale for Practicing Pelvic Floor Exercises (SESPPFE) | At baseline in both groups. Participants in the intervention group will also be asked to answer the questionnaire again within the first month of the intervention period
  The participants will be asked to rate their self-efficacy (from 0-100) on 16 different items regarding PFM training. The scale have been tested to have good internal consistency (α = 0.92) and acceptable reliability (rho = 0.89).
Anal incontinence | Change in score from baseline at four months
  Questions from patient-reported outcome measures (PROM) with Grade A recommendation from the International Consensus on Incontinence 2017 will be used to assess prevalence and bother of anal incontinence (ICIQ-B)
Pelvic Organ Prolapse | Change in score from baseline at four months
  Questions from patient-reported outcome measures (PROM) with Grade A recommendation from the International Consensus on Incontinence 2017 will be used to assess prevalence and bother of pelvic organ prolapse (ICIQ-VS).
Patient Global Impression of Improvement (PGI-I) Scale | Post-test after a 4-months intervention period
  The participants will be asked to rate their perceived change of the condition. A validated 7-point scale with response choices ranging from "very much better" to "very much worse" will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Bø, PhD, Study Chair — Norwegian School of School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Department of Sport Medicine, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piercy KL, Troiano RP. Physical Activity Guidelines for Americans From the US Department of Health and Human Services. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e005263. doi: 10.1161/CIRCOUTCOMES.118.005263. No abstract available. PMID 30571339
- [Background] Ruiz-Zapata, A. M., Feola, A. J., Heesakkers, J., de Graaf, P., Blaganje, M., & Sievert, K. D. (2018). Biomechanical Properties of the Pelvic Floor and its Relation to Pelvic Floor Disorders. European Urology Supplements, 17(3), 80-90.
- [Background] Bump RC, Norton PA. Epidemiology and natural history of pelvic floor dysfunction. Obstet Gynecol Clin North Am. 1998 Dec;25(4):723-46. doi: 10.1016/s0889-8545(05)70039-5. PMID 9921553
- [Background] Milsom, I., Altman, D., Cartwright, R., Lapitan, M. C. M., Nelson, R., Sjöström, S., & Tikkinen, K. A. O. (2017). Epidemiology of urinary incontinence (UI) and other lower urinary tract symptoms (LUTS), pelvic organ prolapse (POP) and anal (AI) incontinence. In P. C. Abrams, L.; Wagg, A.; Wein, A. (Ed.), Incontinence (Vol. 1, pp. 1-141). Tokyo: 6th International Consultation on Incontinence.
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Bø, K. (2015). Pelvic floor dysfunction, prevention and treatment in elite athletes. In K. Bø, B. Berghmans, S. Mørkved, & M. Van Kampen (Eds.), Evidence based Physical Therapy for the Pelvic Floor - Bridging science and clinical practice (pp. 397-407). Edinburgh London New York Oxford Philadelphia St Louis Sydney Toronto: Elsevier Churchilll Livingstone.
- [Background] de Mattos Lourenco TR, Matsuoka PK, Baracat EC, Haddad JM. Urinary incontinence in female athletes: a systematic review. Int Urogynecol J. 2018 Dec;29(12):1757-1763. doi: 10.1007/s00192-018-3629-z. Epub 2018 Mar 19. PMID 29552736
- [Background] Nygaard IE, Shaw JM. Physical activity and the pelvic floor. Am J Obstet Gynecol. 2016 Feb;214(2):164-171. doi: 10.1016/j.ajog.2015.08.067. Epub 2015 Sep 6. PMID 26348380
- [Background] Jacome C, Oliveira D, Marques A, Sa-Couto P. Prevalence and impact of urinary incontinence among female athletes. Int J Gynaecol Obstet. 2011 Jul;114(1):60-3. doi: 10.1016/j.ijgo.2011.02.004. Epub 2011 May 14. PMID 21571270
- [Background] Nygaard IE, Thompson FL, Svengalis SL, Albright JP. Urinary incontinence in elite nulliparous athletes. Obstet Gynecol. 1994 Aug;84(2):183-7. PMID 8041527
- [Background] Poswiata A, Socha T, Opara J. Prevalence of stress urinary incontinence in elite female endurance athletes. J Hum Kinet. 2014 Dec 30;44:91-6. doi: 10.2478/hukin-2014-0114. eCollection 2014 Dec 9. PMID 25713669
- [Background] Eliasson K, Edner A, Mattsson E. Urinary incontinence in very young and mostly nulliparous women with a history of regular organised high-impact trampoline training: occurrence and risk factors. Int Urogynecol J Pelvic Floor Dysfunct. 2008 May;19(5):687-96. doi: 10.1007/s00192-007-0508-4. Epub 2008 Jan 26. PMID 18224267
- [Background] Skaug KL, Engh ME, Frawley H, Bo K. Prevalence of Pelvic Floor Dysfunction, Bother, and Risk Factors and Knowledge of the Pelvic Floor Muscles in Norwegian Male and Female Powerlifters and Olympic Weightlifters. J Strength Cond Res. 2022 Oct 1;36(10):2800-2807. doi: 10.1519/JSC.0000000000003919. Epub 2020 Dec 3. PMID 33278274
- [Background] Wikander L, Kirshbaum MN, Waheed N, Gahreman DE. Urinary Incontinence in Competitive Women Powerlifters: A Cross-Sectional Survey. Sports Med Open. 2021 Dec 7;7(1):89. doi: 10.1186/s40798-021-00387-7. PMID 34874496
- [Background] Wikander L, Kirshbaum MN, Waheed N, Gahreman DE. Urinary Incontinence in Competitive Women Weightlifters. J Strength Cond Res. 2022 Nov 1;36(11):3130-3135. doi: 10.1519/JSC.0000000000004052. Epub 2021 Jun 3. PMID 34100787
- [Background] Elks W, Jaramillo-Huff A, Barnes KL, Petersen TR, Komesu YM. The Stress Urinary Incontinence in CrossFit (SUCCeSS) Study. Female Pelvic Med Reconstr Surg. 2020 Feb;26(2):101-106. doi: 10.1097/SPV.0000000000000815. PMID 31990796
- [Background] Forner LB, Beckman EM, Smith MD. Do women runners report more pelvic floor symptoms than women in CrossFit(R)? A cross-sectional survey. Int Urogynecol J. 2021 Feb;32(2):295-302. doi: 10.1007/s00192-020-04531-x. Epub 2020 Sep 21. PMID 32955598
- [Background] Poli de Araujo M, Brito LGO, Rossi F, Garbiere ML, Vilela ME, Bittencourt VF; Cross Continence Brazil Collaboration Group. Prevalence of Female Urinary Incontinence in Crossfit Practitioners and Associated Factors: An Internet Population-Based Survey. Female Pelvic Med Reconstr Surg. 2020 Feb;26(2):97-100. doi: 10.1097/SPV.0000000000000823. PMID 31990795
- [Background] Wikander L, Kirshbaum MN, Gahreman DE. Urinary Incontinence and Women CrossFit Competitors. Int J Womens Health. 2020 Dec 14;12:1189-1195. doi: 10.2147/IJWH.S278222. eCollection 2020. PMID 33363412
- [Background] Yang J, Cheng JW, Wagner H, Lohman E, Yang SH, Krishingner GA, Trofimova A, Alsyouf M, Staack A. The effect of high impact crossfit exercises on stress urinary incontinence in physically active women. Neurourol Urodyn. 2019 Feb;38(2):749-756. doi: 10.1002/nau.23912. Epub 2019 Jan 8. PMID 30620148
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Woodley SJ, Boyle R, Cody JD, Morkved S, Hay-Smith EJC. Pelvic floor muscle training for prevention and treatment of urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2017 Dec 22;12(12):CD007471. doi: 10.1002/14651858.CD007471.pub3. PMID 29271473
- [Background] Da Roza T, Brandao S, Mascarenhas T, Jorge RN, Duarte JA. Volume of training and the ranking level are associated with the leakage of urine in young female trampolinists. Clin J Sport Med. 2015 May;25(3):270-5. doi: 10.1097/JSM.0000000000000129. PMID 25010151
- [Background] Rivalta M, Sighinolfi MC, Micali S, De Stefani S, Torcasio F, Bianchi G. Urinary incontinence and sport: first and preliminary experience with a combined pelvic floor rehabilitation program in three female athletes. Health Care Women Int. 2010 May;31(5):435-43. doi: 10.1080/07399330903324254. PMID 20390664
- [Background] Sherman RA, Davis GD, Wong MF. Behavioral treatment of exercise-induced urinary incontinence among female soldiers. Mil Med. 1997 Oct;162(10):690-4. PMID 9339085
- [Background] Ferreira, S., Ferreira, M., Carvalhais, A., Santos, P. C., Rocha, P., & Brochado, G. (2014). Reeducation of pelvic floor muscles in volleyball athletes. Rev Assoc Med Bras, 60(5), 428-433.
- [Background] Morkved S, Bo K. The effect of postpartum pelvic floor muscle exercise in the prevention and treatment of urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1997;8(4):217-22. doi: 10.1007/BF02765817. PMID 9449300
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Braekken IH, Stuge B, Tveter AT, Bo K. Reliability, validity and responsiveness of pelvic floor muscle surface electromyography and manometry. Int Urogynecol J. 2021 Dec;32(12):3267-3274. doi: 10.1007/s00192-021-04881-0. Epub 2021 Jun 17. PMID 34142181
- [Background] Tennfjord MK, Engh ME, Bo K. An intra- and interrater reliability and agreement study of vaginal resting pressure, pelvic floor muscle strength, and muscular endurance using a manometer. Int Urogynecol J. 2017 Oct;28(10):1507-1514. doi: 10.1007/s00192-017-3290-y. Epub 2017 Mar 16. PMID 28299404
- [Background] Bø, K. (1992). Pressure measurements during pelvic floor muscle contractions: the effect of different positions of the vaginal measuring device. Neurourol Urodyn, 11, 107-113.
- [Background] Bø, K., Kvarstein, B., Hagen, R., & Larsen, S. (1990a). Pelvic floor muscle exercise for the treatment of female stress urinary incontinence: II.Validity of vaginal pressure measurements of pelvic floor muscle strength and the necessity of supplementary methods for control of correct contraction. Neurourol Urodyn, 9, 479-487.
- [Background] Nystrom E, Sjostrom M, Stenlund H, Samuelsson E. ICIQ symptom and quality of life instruments measure clinically relevant improvements in women with stress urinary incontinence. Neurourol Urodyn. 2015 Nov;34(8):747-51. doi: 10.1002/nau.22657. Epub 2014 Aug 22. PMID 25154378
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Sacomori C, Cardoso FL, Porto IP, Negri NB. The development and psychometric evaluation of a self-efficacy scale for practicing pelvic floor exercises. Braz J Phys Ther. 2013 Jul-Aug;17(4):336-42. doi: 10.1590/S1413-35552013005000104. Epub 2013 Aug 30. English, Portuguese. PMID 24072223
- [Background] Diaz, D. C., Robinson, D., Bosch, R., Constantini, E., Cotterill, N., Espuna-Pons, M., . . . Yoshida, M. (2017). Patient-reported outcome assessment. In P. Abrams, L. Cardozo, A. Wagg, & A. Wein (Eds.), Incontinence (6 ed., Vol. 1, pp. 541-598). Tokyo: 6th International Consultation on Incontinence.